CLINICAL TRIAL: NCT02184156
Title: A Prospective Phase 1/2 Study to Evaluate the Safety and Exploratory Efficacy of Three Intra-articular Injections of Ampion™ (4 mL) Administered Two Weeks Apart in Adults With Pain Due to Osteoarthritis of the Knee
Brief Title: A Study to Evaluate Safety of Three Intra-articular Injections of Ampion in the Knee of Adults With Osteoarthritis Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ampio Pharmaceuticals. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-007
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Results first posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMPION™ 4 mL dose (Experimental): 4 mL injection of Ampion
  Interventions: Biological: 4 mL injection of Ampion
- Placebo 4 mL dose (Placebo Comparator): 4 mL injection of placebo
  Interventions: Drug: 4 mL injection of Placebo

INTERVENTIONS:
Biological: 4 mL injection of Ampion — 4 mL injection of Ampion
  Arms: AMPION™ 4 mL dose
Drug: 4 mL injection of Placebo
  Other Names: Saline
  Arms: Placebo 4 mL dose

SUMMARY:
Phase 1 will evaluate the safety of 3 intra-articular injections of Ampion™ administered 2 weeks apart to adults with osteoarthritis of the knee.

In the absence of serious drug-related Adverse Events (AEs) of unanticipated drug-related AEs, enrollment will be initiated in Phase 2 of the study.

Phase 2 will evaluate the efficacy of 3 intra-articular injections, given 2 weeks apart, of Ampion™ in Adults with pain due to osteoarthritis of the knee.

DETAILED DESCRIPTION:
Phase 1: An open-label study to evaluate the safety of 3 intra-articular injections of of Ampion™ 4 mL at Baseline (Day 0) and Weeks 2 and 4 to adults with osteoarthritis (OA) knee pain. Enrollment will be initiated in Phase 2 if no serious drug-related adverse events or unanticipated drug-related adverse events are observed.

Phase 2: A randomized, placebo-controlled, double-blind, study to evaluate the safety and efficacy of 3 intra-articular (IA) injections of Ampion™ 4 mL at Baseline (Day 0) and Weeks 2 and 4 in adults with OA knee pain.

Study Objectives

Phase 1:

To evaluate the safety of Ampion™ 4 mL administered as 3 intra-articular injections, two weeks apart, in subjects suffering from OA of the knee from Baseline to Week 20.

Phase 2:

The primary study objective is to evaluate the safety and efficacy of Ampion™ 4 mL versus placebo injection from Baseline to Week 20, when administered as three intra-articular (IA) injections (at Baseline (Day 0) and Weeks 2 and 4), in improving knee pain in subjects suffering from OA of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent to participate in the study
2. Willing and able to comply with all study requirements and instructions of the site study staff
3. Male or female, 40 years to 85 years old (inclusive)
4. Ambulatory
5. Index knee must have been symptomatic for greater than 6 months with a clinical diagnosis of OA and supported by radiological evidence (Kellgren Lawrence Grade II-IV) acquired at Screening
6. Moderate to moderately severe OA pain in the index knee (rating of at least 1.5 on the WOMAC Pain Subscale) assessed at Screening and confirmed at randomization
7. Moderate to moderately severe OA pain in the index knee (even if chronic doses of nonsteroidal anti-inflammatory drugs [NSAIDs], which have not changed in the 4 weeks prior to Screening, had been used)
8. No analgesia taken 24 hours before efficacy measure

Exclusion Criteria:

1. As a result of medical review and screening investigation, the Principal Investigator considered the subject unfit for the study
2. Previous Ampion injection
3. Known clinically significant liver abnormality (eg, cirrhosis, transplant, etc.)
4. History of allergic reactions to human albumin (reaction to non-human albumin such as egg albumin was not an exclusion criterion)
5. History of allergic reactions to excipients in 5% human albumin (N-acetyltryptophan, sodium caprylate)
6. Presence of tense effusions in the index knee
7. Inflammatory or crystal arthropathies, acute fractures, history of aseptic necrosis or joint replacement in the index knee, as assessed locally by the Principal Investigator
8. Isolated patella femoral syndrome, also known as chondromalacia in the index knee
9. Any other disease or condition interfering with the free use and evaluation of the index knee for the duration of the trial (eg, cancer, congenital defects, spine OA)
10. Major injury to the index knee within the 12 months prior to Screening
11. Severe hip OA ipsilateral to the index knee
12. Any pain that could interfere with the assessment of index knee pain (eg, pain in any other part of the lower extremities, pain radiating to the knee)
13. Any pharmacological or non-pharmacological treatment targeting OA started or changed during the 4 weeks prior to treatment or likely to be changed during the duration of the study
14. Use of any of the following medications:

    * IA-injected pain medications in the index knee during the study
    * Analgesics containing opioids (NSAIDs were allowed at the levels preceding the study and acetaminophen was available as rescue medication during the study from the provided supply)
    * Topical prescription treatment on the index knee during the study
    * Significant anticoagulant therapy (eg, heparin or enoxaparin) during the study (aspirin and clopidogrel were allowed)
    * Systemic treatments that could interfere with safety or efficacy assessments during the study
    * Immunosuppressants
    * Corticosteroids >10 mg prednisolone equivalent per day or corticosteroids at doses ≤10 mg prednisolone equivalent that had been changed during the study
15. Any human albumin treatment in the 3 months before randomization

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, M.D., Study Director — Ampio Pharmaceuticals. Inc.
Locations (1):
- Ampio Pharmaceuticals, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schwappach J, Dryden SM, Salottolo KM. Preliminary Trial of Intra-articular LMWF-5A for Osteoarthritis of the Knee. Orthopedics. 2017 Jan 1;40(1):e49-e53. doi: 10.3928/01477447-20160926-02. Epub 2016 Sep 30. PMID 27684085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of subjects for Phase 1 occurred in June and July 2014. Recruitment for Phase 2 occurred in medical clinics during the months of August, September, and October 2014.
Pre-assignment Details: No pharmacological or non-pharmacological treatment targeting osteoarthritis (OA) started or changed during the 4 weeks prior to randomization or likely to be changed during the duration of the study.
Groups:
- Ampion 4mL: 4 mL intra-articular injection of Ampion
  Ampion <5 kDa ultrafiltrate of 5% human serum albumin: 4 mL intra-articular injection of Ampion
- Placebo 4 mL: 4 mL placebo intra-articular injection
  Placebo: Saline
Period: Phase 1 Safety
Arm/Group | Ampion 4mL | Placebo 4 mL
Started | 7 | 0
Completed | 7 | 0
Not Completed | 0 | 0
Period: Phase 2 20 Week Efficacy
Arm/Group | Ampion 4mL | Placebo 4 mL
Started | 20 | 20
Completed | 19 | 19
Not Completed | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1 Safety Study Population; Phase 2 20 Week Efficacy Population
Groups:
- Phase 1 - Ampion 4 mL Injection: Non-Randomized; 4 mL Intra-articular injection of Ampion
- Phase 2 - Ampion 4 mL Injection: 4 mL Intra-articular injection of Ampion
- Phase 2 - Placebo 4 mL Injection: 4 mL placebo intra-articular injection
  Placebo: Saline
- Total: Total of all reporting groups
Arm/Group | Phase 1 - Ampion 4 mL Injection | Phase 2 - Ampion 4 mL Injection | Phase 2 - Placebo 4 mL Injection | Total
Number analyzed (Participants) | 7 | 20 | 20 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (9.8) | 63.7 (10.3) | 61.4 (9.4) | 62.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 12 | 13 | 26
  Male | 6 | 8 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 7 | 18 | 19 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 17 | 20 | 44
  More than one race | 0 | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 20 | 20 | 47
Kellgren-Lawrence (KL) Grade [Count of Participants; unit: Participants] — Kellgren-Lawrence grading is based on the radiologic features of osteoarthritis.
  Ann Rheum Dis. 1957;16:494-502. Grade II (Mild): Definite osteophytes, possible joint space narrowing. Grade III (Moderate): Moderate osteophytes, definite joint space narrowing, some sclerosis, possible bone-end deformity.
  Grade IV (Severe): Large osteophytes, marked joint space narrowing, severe sclerosis, definite bone-end deformity
  Participants
    Kellgren-Lawrence Grade II | 0 | 2 | 0 | 2
    Kellgren-Lawrence Grade III | 4 | 11 | 12 | 27
    Kellgren-Lawrence Grade IV | 3 | 7 | 8 | 18
Weight [Mean (Standard Deviation); unit: Pounds] | 188.9 (35.2) | 197.6 (44.7) | 193.8 (44.4) | 194.7 (42.5)
BMI [Mean (Standard Deviation); unit: lbs/in^2] | 27.2 (4.6) | 29.8 (5.1) | 29.9 (4.9) | 29.5 (4.9)
WOMAC Pain [Mean (Standard Deviation); unit: score on a scale] — The Western Ontario and McMaster Universities Arthritis Index (WOMAC) 3.1 evaluates Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright.
  Subjects respond to each subscale by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme). Mean of the 5 scores constitutes the Baseline Pain Score. The minimum score on this scale is 0, and the maximum score is 4. Higher scores are indicative of higher levels of self-reported pain. Population: Phase 1 was a safety study that did not study efficacy. Thus, this baseline measure was not collected.
  score on a scale
    number analyzed (Participants) | 0 | 20 | 20 | 40
    (all) |  | 2.23 (0.47) | 2.17 (0.44) | 2.21 (0.46)
WOMAC Function [Mean (Standard Deviation); unit: score on a scale] — WOMAC 3.1 evaluates Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, rising from bed, lying in bed, getting in/out of bath, sitting, getting on/off toilet, heavy/light domestic duties.
  Subjects respond to each by using a 5-point Likert score. (0=none; 1=mild; 2=moderate; 3=severe; 4=extreme).
  Mean of the 17 scores constitutes the Baseline Function Score. Minimum score is 0; maximum is 4.
  Higher scores indicate of higher levels of limitations of self-reported physical function. Population: Phase 1 was a safety study that did not study efficacy. Thus, this baseline measure was not collected.
  score on a scale
    number analyzed (Participants) | 0 | 20 | 20 | 40
    (all) |  | 2.17 (0.50) | 2.30 (0.52) | 2.24 (0.51)

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events and Serious Adverse Events (Phase 1)
Description: Incidence and severity of adverse events and serious adverse events evaluated at 24 weeks
Time Frame: 24 Weeks
Population: Safety Population
Measure: Number; unit: events
Units Other Than Participants: events
Arm/Group | Phase 1 - Ampion 4 mL Injection
Number analyzed (Participants) | 7
Number analyzed (events) | 15
events
  Serious Adverse Event | 0
  Any Adverse Event | 15

2. Primary Outcome: Change in Knee Pain (Phase 2)
Description: Mean Change in WOMAC A Pain (Western Ontario and McMaster Universities Arthritis Index) score from Baseline to 12 weeks. 5-point Likert scale (0=none to 4=extreme). A negative difference constitutes a decrease in pain with a greater negative value indicating a greater reduction in pain.
Time Frame: Scored at Baseline and 20 Weeks
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ampion 4 mL Injection: 4 mL Intra-articular injection of Ampion
  Ampion: <5 kilodalton (kDa) ultrafiltrate of 5% human serum albumin
- Placebo 4 mL Injection: 4 mL placebo intra-articular injection
  Placebo: Saline
Arm/Group | Ampion 4 mL Injection | Placebo 4 mL Injection
Number analyzed (Participants) | 20 | 20
score on a scale | -1.41 (0.81) | -0.85 (0.64)
Statistical Analysis 1: Comparison: Ampion 4 mL Injection vs Placebo 4 mL Injection; Test type: Superiority; p = 0.02, t-test, 2 sided

3. Secondary Outcome: Change in Knee Function (Phase 2)
Description: Mean change in WOMAC C function score (Western Ontario and McMaster Universities Arthritis Index) from Baseline to 12 weeks. 5-point Likert scale indicating limitation of function (0=none to 4=extreme). A greater negative value indicates a improvement in function.
Time Frame: Scored at Baseline and 20 Weeks
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Ampion < 5 kDa Ultrafiltrate of 5% HSA: 4 mL intra-articular injection of Ampion
  Ampion <5 kDa ultrafiltrate of 5% human serum albumin: 4 mL intra-articular injection of Ampion
- Placebo Solution: 4 mL placebo intra-articular injection
  Placebo: Saline
Arm/Group | Ampion < 5 kDa Ultrafiltrate of 5% HSA | Placebo Solution
Number analyzed (Participants) | 20 | 20
score on a scale | -1.27 (0.81) | -0.98 (0.69)
Statistical Analysis 1: Comparison: Ampion < 5 kDa Ultrafiltrate of 5% HSA vs Placebo Solution; Test type: Superiority; p = 0.25, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 Weeks
Description: Patients will be followed for the occurrence of Adverse Events until 24 weeks after the first dose of study medication
Groups:
- Ampion 4 mL (Phase 1): Non-Randomized; 4 mL Intra-articular injection of Ampion
- Ampion 4 mL (Phase 2): 4 mL intra-articular injection of Ampion
  Ampion <5 kDa ultrafiltrate of 5% human serum albumin: 4 mL intra-articular injection of Ampion
- Placebo 4 mL (Phase 2): 4 mL placebo intra-articular injection
  Placebo: Saline
Arm/Group | Ampion 4 mL (Phase 1) | Ampion 4 mL (Phase 2) | Placebo 4 mL (Phase 2)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/7 | 3/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/7 | 19/20 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ampion 4 mL (Phase 1) (N=7) | Ampion 4 mL (Phase 2) (N=20) | Placebo 4 mL (Phase 2) (N=20)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ampion 4 mL (Phase 1) (N=7) | Ampion 4 mL (Phase 2) (N=20) | Placebo 4 mL (Phase 2) (N=20)
Vision Blurred (Eye disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Injection Site Discolouration (General disorders) | 0 | 2 | 0
Injection Site Haematoma (General disorders) | 0 | 3 | 0
Injection Site Joint Pain (General disorders) | 0 | 1 | 0
Injection Site Pain (General disorders) | 1 | 1 | 3
Oedema Peripheral (General disorders) | 0 | 2 | 0
Vessel Puncture Site Haematoma (General disorders) | 0 | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 1 | 0
Pertussis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1
Back Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 2 | 1
Joint Injury (Injury, poisoning and procedural complications) | 1 | 4 | 2
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural Site Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 1 | 0 | 0
Neck injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The Phase 2 study was underpowered to detect a statistically significant change in function.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes